**Date:** 25/01/2022

Official Title: The Effect of Different Neuromodulation Techniques

in the Treatment of Multiple Sclerosis Patients With Neurogenic

Bladder Dysfunction

## **Statistical Analysis Plan**

Statistical analysis of the data obtained from the study will be done in the SPSS 22.0 package program. The mean standard deviation, median, minimum and maximum values will be used to define the data. Comparison of continuous variables between groups will be done with Mann Whitney U test, comparison of discrete variables will be done with chi-square test. Spearman or Pearson correlation test will be used to evaluate the correlation between variables. In the data analysis, p < 0.05 level will be considered statistically significant.